CLINICAL TRIAL: NCT05290480
Title: Expiratory Muscle Training Versus Incentive Spirometry After Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erhan KIZMAZ, research assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ekizmaz
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer; Pulmonary Rehabilitation
Keywords: Colorectal surgery; Expiratory muscle training; Pulmonary rehabilitation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Treatment and evaluation were performed by two different physiotherapists. The assessing physiotherapist was blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expiratory muscle training (Experimental): participant performed expiratory muscle training with threshold device
  Interventions: Other: expiratory muscle training
- Insentive spirometry (Experimental): participant performed deep breathing exercise with insentive spirometry device
  Interventions: Device: Insentive spirometry

INTERVENTIONS:
Other: expiratory muscle training — participants performed expiratory muscle training according to their maximum expiratory pressure that measured earlier in addition to conventional chest physiotherapy
  Arms: Expiratory muscle training
Device: Insentive spirometry — participants performed deep breating exercise with insentive spirometry in additional to convantional chest physiotherapy
  Arms: Insentive spirometry

SUMMARY:
The aim of this study was to compare the effects of expiratory muscle training (EMT) and incentive spirometry (IS) in addition to conventional pulmonary rehabilitation after colorectal surgery. Twenty-four individuals (13 male) undergoing colorectal surgery were included. They were randomly divided into two groups. In addition to conventional chest physiotherapy, group 1 was performed EMT (n=12), group 2 was performed deep breathing exercises with incentive spirometry (IS) in postoperative period. Respiratory muscle strength, functional capacity, levels of movement and independence, and postoperative pulmonary complications (PPC) were evaluated. Length of stay in hospital (LOS) was recorded.

DETAILED DESCRIPTION:
The aim of this study was to compare the effects of expiratory muscle training (EMT) and incentive spirometry (IS) in addition to conventional pulmonary rehabilitation after colorectal surgery. Twenty-four individuals (13 male) undergoing colorectal surgery were included. They were randomly divided into two groups. In addition to conventional chest physiotherapy, group 1 was performed EMT (n=12), group 2 was performed deep breathing exercises with incentive spirometry (IS) in postoperative period. Respiratory muscle strength, functional capacity, levels of movement and independence, and postoperative pulmonary complications (PPC) were evaluated. Length of stay in hospital (LOS) was recorded

ELIGIBILITY:
Inclusion Criteria:

* hemodynamically stable
* able to walk independently
* able to walk independently

Exclusion Criteria:

* any contraindication for chest physiotherapy (unstable cardiovascular disease, severe pulmonary hypertension, corrected severe hypoxemia, exercise desaturation, rib fractures, subcutaneous emphysema, advanced osteoporosis, thrombocytopenia, effort dyspnea and vertigo)
* any metastases
* severe chronic cardiovascular disease
* candidates for organ transplantation
* abdominal hernia repair
* history of surgery more than one year
* orthopaedic or neurological disease that would prevent independent walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | 2-3 minutes
  Maximum expiratory and inspiratory muscle strength
Postoperative pulmonary complications | 3-7 day
  any pulmonary complications after colorectal surgery
6 Minutes walk test | 6-10 minutes
  Physical functional capacity
'Patient Mobility and Observer Mobility Scale | 2-3 days
  Indipendence and mobility levels after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Erhan KIZMAZ, Msc, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No